CLINICAL TRIAL: NCT02633371
Title: A Pilot Study Exploring the Efficacy and Safety of Topical Oxybutynin 3% Gel for Primary Focal Hyperhidrosis in Adolescents and Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0847; UL1TR001082 (NIH)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxybutynin (Experimental): Oxybutynin 3% gel, 1 gram of product (56 mg oxybutynin) topically to each armpit daily for 4 weeks
  Interventions: Drug: Oxybutynin 3% gel

INTERVENTIONS:
Drug: Oxybutynin 3% gel
  Other Names: Gelnique

SUMMARY:
This is a single-center, prospective, open-label, outpatient pilot study evaluating the efficacy and tolerability of oxybutynin gel for axillary hyperhidrosis.

DETAILED DESCRIPTION:
This study will determine if daily application of topical oxybutynin 3% gel reduces the symptoms of primary axillary hyperhidrosis in adolescents and young adults. It will also assess the impact of daily topical oxybutynin 3% gel on Health Related Quality of Life (HRQOL); determine if daily topical oxybutynin 3% gel has a treatment effect at distant, untreated sites; and assess the local and systemic tolerability of daily topical oxybutynin 3% gel. Finally, the study will determine the treatment effect size, if one exists, in order to power a larger, placebo-controlled study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must be 12-25 years old and meet consensus criteria for primary focal hyperhidrosis: focal, visible, excessive sweating of at least 6 months duration without apparent cause with at least two of the following characteristics: 1) Bilateral and relatively symmetric, 2) Impairs daily activities, 3) Frequency of at least one episode per week, 4) Age of onset less than 25 years, 5) Positive family history, 6) Cessation of focal sweating during sleep.
* Eligible subjects must have moderate to severe hyperhidrosis which correlates to a score of 3 or 4 on the HDSS.
* Hyperhidrosis must affect the bilateral axilla; however, patients with concurrent focal hyperhidrosis affecting the palms, soles, face, or other area will not be excluded.
* Subjects must be willing to comply with the study protocol.

Exclusion Criteria:

* Subjects with hyperhidrosis of less than 6 months duration or hyperhidrosis secondary to an underlying infectious, endocrine, or neurologic disorder.
* Treatment with botulinum toxin injections to the axillae or other affected areas within the last 12 weeks OR treatment with other agents (oral anticholinergic medications, topical aluminum chloride) in the last 4 weeks.
* Subjects with active skin inflammation or infection affecting the axilla
* Subjects who report history of closed-angle glaucoma, urinary retention, decreased gastrointestinal motility, hiatal hernia, cardiac arrhythmia, coronary artery disease, congestive health failure, hyperthyroidism, myasthenia gravis, xerostomia, renal insufficiency, or hepatic impairment.
* Subjects with hypertension defined as systolic blood pressure > 140 or diastolic blood pressure > 90 on more than 1 occasion separated by 1 week.
* Subjects with the following: history of somnolence, confusion, hallucinations OR subjects taking other medications that may cause somnolence, confusion, hallucinations OR subjects with other medical conditions that may predispose them for somnolence, confusion, or hallucinations.
* Subjects who have demonstrated hypersensitivity to the drug substance or other components of the product
* Subjects taking drugs which inhibit Cytochrome P450 3A4 (CYP3A4)
* Pregnant and/or nursing females
* Any other disease that would interfere with the study or place them at undue risk or who are in any way unable to comply with study requirements.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna L Bruckner, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital, Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxybutynin
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Oxybutynin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 18.5 [13 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improvement in Hyperhidrosis Severity at Week 1 or Week 4 as Measured by the Hyperhidrosis Disease Severity Scale (HDSS).
Description: A treatment responder is defined as any participant with a change in the Hyperhidrosis Disease Severity Scale (HDSS) score from a baseline score of 3 or 4 to a score of 1 or 2 at week 1 or week 4.
Time Frame: Week 1 and week 4
Measure: Number; unit: participants
Arm/Group | Oxybutynin
Number analyzed (Participants) | 7
participants | 4

ADVERSE EVENTS:
Groups:
- Oxybutynin: Oxybutynin 3% gel, 1 gram of product (56 mg oxybutynin) topically to each armpit daily for 4 weeks
  Oxybutynin 3% gel
Arm/Group | Oxybutynin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin (N=10)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin (N=10)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Blurry vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No